CLINICAL TRIAL: NCT01062061
Title: Re-examination Study for General Vaccine Use to Assess the Safety Profile of Varivax in Usual Practice
Brief Title: Re-examination Study For Varivax (V210-059 AM2)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: V210-059; 2010_004 (Other: Merck)
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Results first posted 2013-07-03 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Varicella
Keywords: Varicella
MeSH Terms: conditions — Chickenpox | interventions — Chickenpox Vaccine

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VARIVAX: Attenuated live varicella vaccine was administered in usual practice. Recommended dosing is a single 0.5 mL subcutaneous injection in children 12 months to 12 years of age.
  Interventions: Biological: VARIVAX™

INTERVENTIONS:
Biological: VARIVAX™ — Attenuated live varicella vaccine

SUMMARY:
This survey is conducted for preparing application materials for re-examination under the Korean Pharmaceutical Affairs Laws and its Enforcement Regulation; its aim is to reconfirm the clinical usefulness of VARIVAX through collecting the safety information according to the Re-examination Regulation for New Drugs.

DETAILED DESCRIPTION:
This post-marketing survey was conducted in the usual routine practice and the investigator enrolled participants vaccinated with VARIVAX continuously after study start. The purpose of the study was to assess the occurrence of adverse events and to identify factors that may affect the safety of the vaccine under real-life, post-marketing conditions. No hypothesis testing was conducted in this survey.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be vaccinated with VARIVAX as a standard of care

Exclusion Criteria:

* Participants who have been previously vaccinated with VARIVAX
* Contraindication with VARIVAX

Min Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Korean participants being vaccinated with VARIVAX in usual practice
Sampling Method: Probability Sample
Enrollment: 754 (Actual)
Dates: Start 2007-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VARIVAX
Started | 754
Completed | 727
Not Completed | 27
Not completed — Enrolled more than once | 2
Not completed — Investigated before study start | 13
Not completed — Outside chief indications | 10
Not completed — Failed to meet inclusion criteria | 2

BASELINE CHARACTERISTICS:
Arm/Group | VARIVAX
Number analyzed (Participants) | 727
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.19 (0.92)
Age, Customized [Number; unit: Participants]
  <2 years | 686
  ≥2 years | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 347
  Male | 380

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With One or More Adverse Events (AEs)
Description: An adverse event is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the study vaccine, is also an adverse event.
  Changes resulting from normal growth and development which do not vary significantly in frequency or severity from expected levels are not to be considered adverse events. Examples of this may include, but are not limited to, teething, typical crying in infants and children, and onset of menses or menopause occurring at a physiologically appropriate time.
Time Frame: Up to 42 days after vaccination
Population: Adverse events were reported for participants in the safety population: participants administered VARIVAX in usual practice and not discontinued for a reason given in the Participant Flow
Measure: Number; unit: Percentage of Participants
Arm/Group | VARIVAX
Number analyzed (Participants) | 727
Percentage of Participants | 37.69

2. Primary Outcome: Percentage of Participants With One or More AEs by Gender
Description: as for outcome 1
Time Frame: Up to 42 days after vaccination
Population: AEs were reported for participants in the safety population: participants administered VARIVAX in usual practice and not discontinued for a reason given in the Participant Flow
Measure: Number; unit: percentage of participants
Groups:
- Male Participants; Female Participants: Attenuated live varicella vaccine was administered in usual practice. Recommended dosing is a single 0.5 mL subcutaneous injection in children 12 months to 12 years of age.
Arm/Group | Male Participants | Female Participants
Number analyzed (Participants) | 380 | 347
percentage of participants | 37.63 | 37.75
Statistical Analysis 1: Comparison: Male Participants vs Female Participants; Test type: Superiority or Other; p = 0.9733, Chi-squared

3. Primary Outcome: Percentage of Participants With One or More AEs by Age
Description: as for outcome 1
Time Frame: Up to 42 days after vaccination
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Groups:
- Age <2 Years; Age ≥2 Years: Attenuated live varicella vaccine was administered in usual practice. Recommended dosing is a single 0.5 mL subcutaneous injection in children 12 months to 12 years of age.
Arm/Group | Age <2 Years | Age ≥2 Years
Number analyzed (Participants) | 686 | 41
percentage of participants | 36.01 | 65.85
Statistical Analysis 1: Comparison: Age <2 Years vs Age ≥2 Years; Test type: Superiority or Other; p = 0.0001, Chi-squared

4. Primary Outcome: Percentage of Participants With One or More Adverse Drug Reactions (ADRs)
Description: An ADR is an AE (defined above) for which relatedness to the use of the product cannot be ruled out
Time Frame: Up to 42 days after vaccination
Population: ADRs were reported for participants in the safety population: participants administered VARIVAX in usual practice and not discontinued for a reason given in the Participant Flow
Measure: Number; unit: percentage of participants
Arm/Group | VARIVAX
Number analyzed (Participants) | 727
percentage of participants | 3.30

5. Primary Outcome: Percentage of Participants With One or More Unexpected AEs
Description: Unexpected AEs differed from AEs reported in the VARIVAX product label with regard to their identity, severity, specificity, or outcome
Time Frame: Up to 42 days after vaccination
Population: Unexpected AEs were reported for participants in the safety population: participants administered VARIVAX in usual practice and not discontinued for a reason given in the Participant Flow
Measure: Number; unit: percentage of participants
Arm/Group | VARIVAX
Number analyzed (Participants) | 727
percentage of participants | 26.00

6. Primary Outcome: Percentage of Participants With One or More Unexpected ADRs
Description: An unexpected ADR is an unexpected AE (defined above) for which relatedness to the use of the study vaccine cannot be ruled out
Time Frame: Up to 42 days after vaccination
Population: Unexpected ADRs were reported for participants in the safety population: participants administered VARIVAX in usual practice and not discontinued for a reason given in the Participant Flow
Measure: Number; unit: percentage of participants
Arm/Group | VARIVAX
Number analyzed (Participants) | 727
percentage of participants | 0.14

7. Primary Outcome: Percentage of Participants With One or More Serious Adverse Events (SAEs)
Description: An SAE is any AE that results in death, is life-threatening, results in persistent or significant disability/incapacity, results in or prolongs an existing inpatient hospitalization, is a congenital anomaly/birth defect, is a cancer, is an overdose, or is another important medical event based on appropriate medical judgment.
Time Frame: Up to 42 days after vaccination
Population: SAEs were reported for participants in the safety population: participants administered VARIVAX in usual practice and not discontinued for a reason given in the Participant Flow
Measure: Number; unit: percentage of participants
Arm/Group | VARIVAX
Number analyzed (Participants) | 727
percentage of participants | 0.55

8. Primary Outcome: Percentage of Participants With One or More Serious ADRs
Description: A serious ADR is an SAE (defined above) for which relatedness to the use of the product cannot be ruled out
Time Frame: Up to 42 days after vaccination
Population: Serious ADRs were reported for participants in the safety population: participants administered VARIVAX in usual practice and not discontinued for a reason given in the Participant Flow
Measure: Number; unit: percentage of participants
Arm/Group | VARIVAX
Number analyzed (Participants) | 727
percentage of participants | 0

9. Primary Outcome: Percentage of Participants With One or More Unexpected SAEs
Description: Unexpected SAEs differed from SAEs reported in the VARIVAX product label with regard to their identity, severity, specificity, or outcome
Time Frame: Up to 42 days after vaccination
Measure: Number; unit: percentage of participants
Arm/Group | VARIVAX
Number analyzed (Participants) | 727
percentage of participants | 0.28

ADVERSE EVENTS:
Time Frame: Up to 42 days after vaccination
Description: Adverse events were reported for participants in the safety population: participants administered VARIVAX in usual practice and not discontinued for a reason given in the Participant Flow
Arm/Group | VARIVAX
Serious Adverse Events (participants affected / at risk) | 4/727
Other Adverse Events (participants affected / at risk) | 105/727
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VARIVAX (N=727)
Pyrexia (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VARIVAX (N=727)
Pyrexia (General disorders) | 51 (59)
Bronchitis (Infections and infestations) | 58 (62)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No